CLINICAL TRIAL: NCT04287400
Title: Prospective Clinical Trial for the Evaluation of Radiogenomics: Correlation, Treatment Response and Prognosis in Patients With Advanced Rectal Cancer, Who Undergo Preoperative Chemoradiation
Brief Title: Prospective Trial for the Evaluation of Radiogenomics in Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, Principal Investigator, National Cancer Center, Korea
Other Study IDs: 2018-0428-0001
Record Dates: First submitted 2019-11-26; First posted 2020-02-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopic cancer biopsy before starting treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients with advanced rectal cancer, molecular subtypes will be identified by preoperative biopsy, CT, MRI / PET radiomics analysis, clinical features, and clinical features will be confirmed and compared.

Also, we want to confirm the relationship between these factors and the treatment response after chemoradiotherapy before surgery. The prognosis will be then assessed through 5-year overall survival and 3-year disease free survival.

A prospective clinical trial, recruiting 210 persons (approximately 53 per year) that meet the selection criteria for approximately four years from the IRB approval date in 2019 (about 53 per year) We will analyze the data and then collect and analyze the data and report the results.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years
* Patients diagnosed with mid-lower rectal cancer and expected to receive chemoradiotherapy before surgery

Exclusion Criteria:

* Patients with distal metastases confirmed at diagnosis
* Patients with other bowel diseases such as IBD, ischemic colitis and TB colitis in addition to colorectal cancer
* If patients do not agree with this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with mid-lower rectal cancer and expected to receive chemoradiotherapy before surgery
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
K-RAS Mutation | 4 weeks
  K-RAS Mutation status

SECONDARY OUTCOMES:
Radiomics - MR image findings | 4 weeks
  Radiologic features

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea